CLINICAL TRIAL: NCT03956134
Title: Investigation of the Pharmacokinetic Characteristics of Two New CG5503 Formulations as Compared to CG5503 PR Tablets and Exploration of the Effect of Food on the Bioavailability of the Two New CG5503 Formulations Following Single Oral Administration of 116 mg CG5503 in a Single Center, Open, Randomized, 5-way-crossover, Single Dose, Phase I Study in 10 Healthy Male Subjects
Brief Title: Pharmacokinetic Characterization of Two Novel CG5503 Tablet Formulations in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Grünenthal GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HP5503/12
Record Dates: First submitted 2019-05-14; First posted 2019-05-20 (Actual); Last update posted 2019-05-20 (Actual); Status verified 2019-05

CONDITIONS: Pharmacokinetics

STUDY DESIGN:
Intervention Model Description: Randomization was performed according to Williams' design, with 5 periods and 10 sequences. There was a washout of at least 3 days between the consecutive administrations.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Tapentadol Test Product 1 (fasting) (Experimental): Tapentadol new tablet formulation, given as single oral dose with 240 mL of still mineral water under fasting condition.
  Interventions: Drug: Tapentadol Test Product 1
- Tapentadol Test Product 2 (fasting) (Experimental): Tapentadol new tablet formulation, given as single oral dose with 240 mL of still mineral water under fasting condition.
  Interventions: Drug: Tapentadol Test Product 2
- Tapentadol Test Product 1 (fed) (Experimental): Tapentadol new tablet formulation, given as single oral dose with 240 mL of still mineral water under fed condition.
  Interventions: Drug: Tapentadol Test Product 1
- Tapentadol Test Product 2 (fed) (Experimental): Tapentadol new tablet formulation, given as single oral dose with 240 mL of still mineral water under fed condition.
  Interventions: Drug: Tapentadol Test Product 2
- Tapentadol PR Reference Product (Active Comparator): Tapentadol PR tablet formulation given as single oral dose with 240 mL of still mineral water under fasting condition.
  Interventions: Drug: Tapentadol Prolonged-release Reference Product

INTERVENTIONS:
Drug: Tapentadol Test Product 1 — Tapentadol tablet containing 116 mg of tapentadol hydrochloride; Tapentadol Test Product 1 contains different amounts of excipients than Tapentadol Test Product 2
  Arms: Tapentadol Test Product 1 (fasting); Tapentadol Test Product 1 (fed)
Drug: Tapentadol Test Product 2 — Tapentadol tablet containing 116 mg of tapentadol hydrochloride; Tapentadol Test Product 2 contains different amounts of excipients than Tapentadol Test Product 1
  Arms: Tapentadol Test Product 2 (fasting); Tapentadol Test Product 2 (fed)
Drug: Tapentadol Prolonged-release Reference Product — Tapentadol PR tablet containing 116 mg of tapentadol hydrochloride
  Arms: Tapentadol PR Reference Product

SUMMARY:
This study investigated the pharmacokinetics (how a drug is taken up and excreted from the body), safety, and tolerability of 2 new tapentadol (CG5503) tablet formulations compared to a previously characterized tapentadol prolonged-release (PR) tablet formulation.

DETAILED DESCRIPTION:
The study was performed to evaluate the pharmacokinetic characteristics (relative bioavailability) of 2 new tapentadol (CG5503) tablet formulations (Test Product 1 and Test Product 2) containing 116 mg tapentadol hydrochloride each, as compared to a 116-mg tapentadol hydrochloride PR tablet (Reference Product) and to explore the effect of food on the bioavailability of the 2 new tapentadol formulations. Participants received a single dose of each of the test formulations under fasting or fed conditions and of the reference formulation under fasting conditions in a randomized order. There was a wash-out period of at least 3 days between consecutive treatments. Blood samples were taken from pre-dose up to 32 hours post-dose for pharmacokinetic analyses.

Furthermore, the study compared the safety and tolerability of the test formulations with that of the reference. Adverse events and vital signs were documented at screening, pre-dose, and up to 32 hours post-dose. Clinical laboratory parameters were determined and 12-lead electrocardiograms (ECG) were recorded at screening and at discharge. A final medical examination was performed at 2-14 days after discharge following the last treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male Caucasian participants, aged 18-55 years;
* Body Mass Index between 18 and 30 kg/m2 inclusive;
* Participants must be in good health as determined by medical history, physical examination, 12-lead electrocardiogram, vital signs, and clinical laboratory parameters;
* Participants giving written informed consent to participate within this study.

Exclusion Criteria:

* Resting pulse rate equal to or less than 45 or equal to or above 95 beats / min;
* Resting blood pressure: systolic blood pressure equal to or less than 100 and equal to or above 140 mmHg, diastolic blood pressure equal to or less than 50 and equal to or above 90 mmHg;
* Positive human immunodeficiency virus (HIV) type 1/2 antibodies, hepatitis B surface (HBs) antigen, hepatitis B core (HBc) antibodies, hepatitis C virus (HCV) antibodies;
* History or presence of orthostatic hypotension;
* Participation in another clinical study in the last three months before starting this study (exception: characterization of metabolizer status);
* Positive screening of drug abuse;
* Diseases or condition known to interfere with the absorption, distribution, metabolism or excretion of drugs;
* Marked repolarization abnormality (e.g., suspicious or definite congenital long QT syndrome);
* Bronchial asthma;
* Definite or suspected history of drug allergy or hypersensitivity;
* Participants who have received any prescribed and non-prescribed systemic or topical medication two weeks before and during the study with the exception of short term medication, e.g. headache with paracetamol;
* Evidence of alcohol or drug abuse;
* Not able to abstain from drinking of caffeine containing beverages (tea, coffee, chocolate or cola),
* Consumption of any quinine containing beverages (bitter lemon, tonic water) or food within two weeks before and during the study;
* Drinking of alcohol containing beverages within 48 hours before administration of investigational product(s);
* Blood donation (above 100 mL) or comparable blood losses during the last 3 months;
* History of seizures or at risk (i.e. head trauma, epilepsy in family anamnesis, unclear loss of consciousness);
* Known or suspected of not being able to comply with the study protocol;
* Not able to communicate meaningfully with the investigator and staff;
* Smoking of more than 20 cigarettes/day.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2005-04 (Actual); Primary Completion 2005-06 (Actual); Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameter: Cmax | Pre-dose up to 32 hours post-dose
  19 Blood samples were collected from pre-dose up to 32 hours post-dose. The evaluation of the maximum observed serum concentration (Cmax) was based on the tapentadol base concentrations measured in serum samples using a validated liquid chromatography/tandem mass spectrometry (LC-MS/MS) method.
Pharmacokinetic parameter: AUC0-t | Pre-dose up to 32 hours post-dose
  19 Blood samples were collected from pre-dose up to 32 hours post-dose. The evaluation of the area under the concentration time curve (AUC) from 0 hours to time t (=32 hours) (AUC0-t) was based on the tapentadol base concentrations measured in serum samples.
Pharmacokinetic parameter: AUC0-inf | Pre-dose up to 32 hours post-dose
  19 Blood samples were collected from pre-dose up to 32 hours post-dose. The AUC from 0 hours to infinity (AUC0-inf) was extrapolated from the AUC from administration to the last measured concentration.
Pharmacokinetic parameter: tmax | Pre-dose up to 32 hours post-dose
  19 Blood samples were collected from pre-dose up to 32 hours post-dose. The evaluation of the time to reach Cmax (tmax) was determined based on the tapentadol base concentrations measured in serum samples.

SECONDARY OUTCOMES:
Pharmacokinetic parameter: MRT | Pre-dose up to 32 hours post-dose
  19 Blood samples were collected from pre-dose up to 32 hours post-dose. The evaluation of the mean residence time (MRT) was based on the tapentadol base concentrations measured in serum samples using a validated LC-MS/MS method.
Pharmacokinetic parameter: CL/f | Pre-dose up to 32 hours post-dose
  19 Blood samples were collected from pre-dose up to 32 hours post-dose. The evaluation of the apparent total clearance from serum after oral administration (CL/f) of tapentadol base was calculated based on available dose and AUC data.
Pharmacokinetic parameter: Vz/f | Pre-dose up to 32 hours post-dose
  19 Blood samples were collected from pre-dose up to 32 hours post-dose. The evaluation of the apparent volume of distribution during the terminal disposition phase (Vz/f) was calculated based on CL/f and terminal elimination rate constant lambda z.
Pharmacokinetic parameter: tlag | Pre-dose up to 32 hours post-dose
  19 Blood samples were collected from pre-dose up to 32 hours post-dose. The evaluation of the lag time (tlag) was based on the tapentadol base concentrations measured in serum samples. Tlag was taken as the time point prior to that of the first quantifiable serum concentration.
Pharmacokinetic parameter: t1/2z | Pre-dose up to 32 hours post-dose
  19 Blood samples were collected from pre-dose up to 32 hours post-dose. The evaluation of the apparent terminal half life (t1/2z) was based on the tapentadol base concentrations measured in serum samples.

CONTACTS AND LOCATIONS:
Overall Officials: Grünenthal Study Director, Study Director — Grünenthal GmbH
Locations (1):
- Department of Clinical Pharmacology, Grünenthal GmbH, Aachen, Germany

IPD SHARING:
Plan to Share IPD: No